CLINICAL TRIAL: NCT05390216
Title: Impact of Partial Capsule Decortication on Device-related Infection in Patients Receiving Cardiac Implantable Electronic Device Replacement: a Multicenter Randomized Controlled Trial
Brief Title: Impact of Partial Capsule Decortication on Device-related Infection in Patients Receiving Cardiac Implantable Electronic Device Replacement
Acronym: STERILE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12901
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pacemaker Complication; Infections
MeSH Terms: conditions — Infections | interventions — Cerebral Decortication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial capsule decortication (Experimental)
  Interventions: Procedure: Partial capsule decortication
- Without partial capsule decortication (No Intervention)

INTERVENTIONS:
Procedure: Partial capsule decortication — The anterior wall of the capsule was removed during the operation.
  Arms: Partial capsule decortication

SUMMARY:
Increasing number of cardiac implantable electronic devices (CIEDs) have been implanted in the worldwide every year, which is accompanied by the growing number of CIED-related infection, especially in patients with CIED replacement. This multicenter, prospective, single-blinded, randomized controlled trial is to confirm the impact of partial capsule decortication on device-related infection in patients receiving CIED replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is planned to undergo at least one of the following procedures:

  a) Patient has existing CIED (pacemaker, or CRT-P, or ICD, or CRT-D) and is undergoing pulse generator replacement or upgrade with a new generator. b) Patients planned to have leads added, or extracted and added for upgrades.
* Patient is willing to sign and date informed consent

Exclusion Criteria:

* History of CIED-related infection
* Open the pocket for any reason within the last one year
* Any evidence indicating active infection
* Requirement of long term vascular access for any reason
* Expected survival time is less than one year
* Patients who were pregnant or breastfeeding
* Participation in another study that may confound the results of this study
* Patient is unable to comply with scheduled follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1016 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of major CIED-related infection | Within the first year after the operation
  Infections that resulted in CIED system removal, an invasive CIED procedure (e.g., pocket revision without removal), treatment with long-term antibiotic therapy (if the patient was not a candidate for system removal) with infection recurrence after discontinuation of antibiotic therapy, or death.

SECONDARY OUTCOMES:
Rate of minor CIED-related infection | Within the first year after the operation
  Infections that do not meet the definition criteria of major CIED infection.
Rate of all CIED-related infection | Within the first year after the operation
  All infections that related to CIED operation.
Rate of pocket hematoma | Within the first year after the operation
  Palpable swelling with fluctuance that extended beyond the device margin but without evidence of infection.
Rate of device dysfunction | Within the first year after the operation
  All the dysfunction of the generators and leads (including abnormal changes of pacing threshold, sensing, impedance, etc.).
All-cause mortality | Within the first year after the operation
  Death regardless of the causes.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No